CLINICAL TRIAL: NCT04399681
Title: The Utility of Bedside Lung Ultrasonography on Diagnosis of COVID-19 at Emergency Department
Brief Title: The Utility of Bedside Lung Ultrasonography on Diagnosis of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ramazan Guven, Professor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KSSEAH--
Record Dates: First submitted 2020-05-21; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: COVID; Pneumonia, Viral
MeSH Terms: conditions — Pneumonia, Viral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suspected COVID-19 Group (Other): Patients who admitted to emergency department with suspicion of COVID 19 pneumonia will be evaluated with POCUS/ bedside lung ultrasound.
  Interventions: Device: Bedside lung ultrasound

INTERVENTIONS:
Device: Bedside lung ultrasound — Point of care ultrasound will be used as bedside lung ultrasound to determine the patients if they have a COVID-19 pneumonia.

SUMMARY:
Novel Coronavirus 2019 Disease (COVID-19) mortality is highly associated with viral pneumonia and its complications. Accurate and prompt diagnosis shown to be effective to improve outcome by providing early treatment strategies. While chest X-ray (CXR) and computerized tomography (CT) are defined as gold standard, given the advantage of being an ionized radiation free, practical technique point of care ultrasound (POCUS) is also reported as a diagnostic tool for COVID-19. There are limited studies regarding the importance of POCUS in diagnosis and review of COVID-19. Therefore the aim of this study is to evaluate the utility of bedside lung ultrasound on diagnosis of COVID-19 for patients admitted to emergency department .

DETAILED DESCRIPTION:
Novel Coronavirus 2019 Disease (COVID-19) mortality is highly associated with viral pneumonia and its complications. Accurate and prompt diagnosis shown to be effective to improve outcome by providing early treatment strategies. While chest X-ray (CXR) and computerized tomography (CT) are defined as gold standard, given the advantage of being an ionized radiation free, practical technique point of care ultrasound (POCUS) is also reported as a diagnostic tool for COVID-19. There are limited studies regarding the importance of POCUS in diagnosis and review of COVID-19. Therefore the aim of this study is to evaluate the utility of bedside lung ultrasound on diagnosis of COVID-19 for patients admitted to emergency department .

ELIGIBILITY:
Inclusion Criteria:

* All patients with an informed consent
* Admission to emergency department with symptoms or signs of COVID-19

Exclusion Criteria:

* Absence of informed consent
* Patients under age of 18
* Presence of acute coronary syndrome
* Presence of chronic lung disease
* Pregnancy
* Presence of trauma
* Patients with a diagnosis of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
Presence of viral pneumonia caused by COVID 19 | 3 months
  Efficacy of POCUS on diagnosis of viral pneumonia caused by COVID 19

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)